CLINICAL TRIAL: NCT06858618
Title: A Phase II Clinical Study to Evaluate the Safety & Tolerability, Antitumor Activity, and Pharmacokinetics of FCN-338 in Combination With Azacitidine or Chemotherapy in Patients With Myeloid Neoplasms
Brief Title: FCN-338 in Combination With Azacitidine or Chemotherapy in Myeloid Neoplasms
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry)
Collaborators: Beijing Fosun Pharmaceutical Technology Development Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCN-338-II201
Record Dates: First submitted 2025-02-04; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-01

CONDITIONS: Safety; Antitumor Activity; PK Profile
Keywords: BCL-2 inhibitor; Acute Myeloid Leukemia; safety; antitumor activity; PK profile
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- relapse/refractory (R/R) AML (Experimental)
  Interventions: Combination Product: FCN-338 + Azacitidine
- 1L fit AML (Experimental)
  Interventions: Combination Product: FCN-338 + erythromycin+ Ara-C

INTERVENTIONS:
Combination Product: FCN-338 + Azacitidine — FCN-338 (400 or 600 mg, PO, QD, D1-28) combined with azacitidine (75mg/m², SC, QD, D1-7), 28 days/cycle
  Arms: relapse/refractory (R/R) AML
Combination Product: FCN-338 + erythromycin+ Ara-C — Induction phase: FCN-338(600 mg, QD, D1-14) , erythromycin (60 mg/m², IV, QD , D1-3) and Ara-C (100 mg/m², IV, QD, D1-7) for 1 to 2 cycles.
  Consolidation phase: FCN-338(600 mg, QD, D1-14) ,Ara-C (1 to 3 g/m²/12h, 6 doses) for 3 to 4 cycles Maintenance phase:FCN-338(600 mg, QD, D1-14) , azacitidine (50 mg/m², SC, QD, D1-5) for the first 12 cycles and FCN-338 (600 mg, QD, D1-14) alone for the rest 12 cycles
  Arms: 1L fit AML

SUMMARY:
This is a Phase 2, open-label, multicenter study to safety & tolerability, antitumor activity, and pharmacokinetics of FCN-338 in Combination with szacitidine (AZA) or chemotherapy(erythromycin, cytarabine(Ara-C)) in Patients with myeloid neoplasms

DETAILED DESCRIPTION:
Primary Objectives:1.To assess the safety and tolerability of FCN-338 in combination with AZA or chemotherapy in patients with myeloid neoplasms. 2. To explore the antitumor activity of FCN-338 combination therapy in patients with myeloid neoplasms.

Secondary Objectives: 1. To assess the pharmacokinetic profile of the FCN-338 combination therapy in patients with myeloid neoplasms.2. To assess the transfusion independence rate in patients with myeloid neoplasms.

There were 2 cohorts based on different combination therapies and different indications.

Cohort A is FCN-338 combined with AZA (75mg/m², SC, QD, D1-7) for the treatment in relapsed/refractory (R/R) acute myeloid leukemia (AML) patients.

Cohort B is FCN-338 combined with intensive chemotherapy for first line (1L) fit AML patients. During the induction phase, patients will be treated with erythromycin (60 mg/m², IV, QD , D1-3) and Ara-C (100 mg/m², IV, QD, D1-7). Patients achieving partial remission (PR) will repeat induction phase once, and patients who do not reach PR after first cycle of induction phase and those who do not achieve complete remission (CR)/Complete remission with incomplete hematological recovery (CRi)/morphologic leukemia-free state (MLFS) after two cycles of induction phase will receive other new antitumor treatments. Patients who achieve CR/CRi/MLFS will undergo consolidation phase with medium- to high-dose Ara-C (1 to 3 g/m²/12h, 6 doses) for 3 to 4 cycles, with the exact dose and number of cycles determined by investigator. Patients with intermediate- to high-risk according to the 2017 European Leukemia Net (ELN) stratification will undergo a total of 24 cycles of maintenance phase after completion of consolidation phase. Maintenance phase will consist of 24 cycles, FCN-338 in combination with AZA (50 mg/m², d1-5) for the first 12 cycles and FCN-338 alone for the rest 12 cycles. FCN-338 will be administered once daily (QD), D1-14 per cycle during induction phase, consolidation phase and maintenance phase.

ELIGIBILITY:
Inclusive Criteria

1. Age ≥18 years.
2. Cohort A: Patients diagnosed with R/RAML (≥5% blasts in the bone marrow) according to the WHO 2016 criteria [excluding acute promyelocytic leukemia (APL) and BCR-ABL positive AML], meeting any of the following definitions:

1) Relapsed AML: Reappearance of leukemic cells in peripheral blood or ≥5% blasts in bone marrow after complete remission (CR, CRi) (excluding other causes such as bone marrow regeneration after consolidation treatment) or infiltration of leukemic cells outside the marrow; 2) Refractory AML: Ineffective after two cycles of standard treatment; Relapsed within 12 months after CR followed by consolidation treatment; Relapsed after 12 months but ineffective with standard chemotherapy; Relapsed two or more times; With persistent extramedullary leukemia.

3. Cohort B: Patients diagnosed with 1L fit AML according to the WHO 2016 criteria [excluding acute promyelocytic leukemia (APL) and BCR-ABL positive AML].

4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2. 5. Expected survival time ≥ 3 months. 6. Adequate bone marrow and organ function. Exclusive Criteria

1. Patients with diagnosis of APL or BCR-ABL-positive AML patients or a history of prior myeloproliferative disease (MPN).
2. With known leukemic infiltration of the central nervous system.
3. Have received allogeneic hematopoietic stem cell transplantation or overt immune cell therapy, or autologous hematopoietic stem cell transplantation within 1 year.
4. Have active fungal, bacterial and/or viral infections including, but not limited to, active Human Immunodeficiency Virus (HIV), viral hepatitis B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLT | At the end of Cycle 1 (each cycle is 28 days)
  Incidence of DLT in DLT observation period
Title: composite CR rate (CRc) | From the first dose to the end of maintenance phase, assessed up to 30 months
  The proportion of CR, CRi and MLFS patients in the efficacy analysis set (EAS)
Minimal residual disease (MRD) negative rate | From the first dose to the end of maintenance phase, assessed up to 30 months
  The proportion of AML patients with CR/CRi/MLFS who were negative for MRD.

SECONDARY OUTCOMES:
Transfusion Independence | From the first dose to the end of maintenance phase, assessed up to 30 months
  The proportion of independence on red blood cell (RBC) and platelet transfusions among those patients who were dependent on RBC and platelet transfusions at baseline.
Time to remission | From the first dose to the first observation of CR/CRi/MLFS, assessed up to 2 months
  Defined as the time from the first dose to the first observation of CR/CRi/MLFS
Event-free survival | From the first dose to induction failure or relapse or death from any cause (whichever occours first), assessed up to 54 months
  Defined as the time from the first dose to induction failure or relapse or death from any cause (whichever occours first).
Duration of remission | From the first observation of CR/CRi/MLFS to tumor progression or death from any cause(whichever occours first), assessed up to 54 months
  Defined as the time from the first observation of CR/CRi/MLFS to tumor progression or death from any cause(whichever occours first).
Overall survival | From the first dose to 30 days after the last dose or the initiation of new antitumor therapy (whichever occours first), assessed up to 30 months
  Defined as the time from the first dose to death from any cause.
Incidence of treatment-emergent adverse events(TEAEs) and treatment-related adverse events (TRAEs) [Safety and Tolerability] | From the first dose to 30 days after the last dose or the initiation of new antitumor therapy (whichever occours first).
  Safety will be evaluated by summarizing DLT, AE, changes in laboratory findings, and changes in vital signs. Adverse events will be summarized for the DLT observation period and the entire treatment period based on the DLT analysis set and the safety analysis set, respectively, and drug-related AEs, SAEs, AEs of toxicity grade ≥3, and AEs leading to discontinuation will be counted. The occurrence of DLT will be assessed specifically for the DLT analysis set.
Cmax of FCN-338 | Up to 24 hours postdose
  Pharmacokinetics of FCN-338 by assesment of the maximum plasma concentration
AUC0-t of FCN-338 | Up to 24 hours postdose
  Pharmacokinetics of FCN-338 by assesment of the Area Under The Plasma Concentration Time Curve From Time 0 To The Time Of The Last Quantifiable Concentration
AUC0-24 of FCN-338 | Up to 24 hours postdose
  Pharmacokinetics of FCN-338 by assesment of the Area Under The Plasma Concentration Time Curve From Time 0 To The 24 hours postdose
AUC0-∞ of FCN-338 | Up to 24 hours postdose
  Pharmacokinetics of FCN-338 by assesment of The Plasma Concentration Time Curve From Time 0 To Infinity
Tmax of FCN-338 | Up to 24 hours postdose
  Pharmacokinetics of FCN-338 by assesment of Time To Maximum Observed Plasma Concentration
t1/2 of FCN-338 | Up to 24 hours postdose
  Pharmacokinetics of FCN-338 by assesment of Terminal Half-life
CL/F of FCN-338 | Up to 24 hours postdose
  Pharmacokinetics of FCN-338 by assesment of Apparent Clearance Of Drug From Plasma After Oral Administration
Vd/F of FCN-338 | Up to 24 hours postdose
  Pharmacokinetics of FCN-338 by assesment of Apparent Volume Of Distribution
Css_max of FCN-338 | Up to 24 hours postdose
  Pharmacokinetics of FCN-338 by assesment of Maximum Observed Plasma Concentration At Steady State
Css_av of FCN-338 | Up to 24 hours postdose
  Pharmacokinetics of FCN-338 by assesment of the Average concentration At Steady State
AUCss of FCN-338 | Up to 24 hours postdose
  Pharmacokinetics of FCN-338 by assesment of the Area Under The Plasma Concentration Time Curve within dosing interval At Steady State
DF of FCN-338 | Up to 24 hours postdose
  Pharmacokinetics of FCN-338 by assesment of fluctuation
MRT | Up to 24 hours postdose
  Pharmacokinetics of FCN-338 by assesment of Mean residence time
Kel of FCN-338 | Up to 24 hours postdose
  Pharmacokinetics of FCN-338 by assesment of the Terminal rate constant.
Css_min of FCN-338 | Up to 24 hours postdose
  Pharmacokinetics of FCN-338 by assesment of Trough Concentration At Steady State

CONTACTS AND LOCATIONS:
Locations (1):
- Union hospital tongjimedical college huzhong university of science and technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: No